CLINICAL TRIAL: NCT02359747
Title: Analysis of Human Genomic DNA in Embryo's Culture Media Targeting on a Single Gene Disease and Point Mutations
Brief Title: Analysis of Human Genomic DNA in Embryo's Culture Media
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cervesi Hospital, Cattolica, Italy (Other)
Responsible Party: Principal Investigator, Palini Simone, Senior Clinica Embryologist Lab Director, Cervesi Hospital, Cattolica, Italy
Other Study IDs: PGD on culture media is easy
Record Dates: First submitted 2015-02-03; First posted 2015-02-10 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Single-Gene Disease
Keywords: free gDNA; culture media
MeSH Terms: interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- In Vitro Fertilization treatment: culture medium discarded after IVF treatment
  Interventions: Genetic: Polymerase Chain Reaction and Whole Genome Amplification

INTERVENTIONS:
Genetic: Polymerase Chain Reaction and Whole Genome Amplification — Polymerase Chain Reaction and Whole Genome Amplification

SUMMARY:
try to find genomic DNA in culture medium after the embryos develop on Day 3 and Day 5 also in single step culture media. using direct PCR Polymerase Chain Reaction and also WGA Whole Genome Amplification before PCR and sequencing of the samples to find the point mutation

DETAILED DESCRIPTION:
Human fertilized oocytes were individually cultured from Day 1 to Day 3, and from day 3 to days 5/6, in 10 ul medium. A total of 100 samples (50 spent media from Day 3 and 50 from Day 5/6) will be use in the study.

Double-stranded DNA (dsDNA) amplifiability will be evaluated in embryos culture media by quantitative PCR on a multicopy gene target (TBC1D3). Quantification will be made with a standard curve constructed with genomic DNA (with culture media -day 3 and day5-, to take into account media inhibitory effects) TSPY1 amplification will be use to assess the presence of Y chromosome WGA followed by PCR on a single copy gene (MTHFR gene) will be performed on a subset of some samples to monitor the C677T polymorphism (genotyping by sequencing) WGA followed by PCR on a single copy gene (MTHFR) will be also performed on blastocoele fluids

ELIGIBILITY:
Inclusion Criteria

* all the patients undergoing IVF treatment at Cervesi Hospital

Exclusion Criteria:

* patients with embryos that can't be cultured from day 0 (insemination day) to day 5/6 (blastocyst stage)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all the mediun descarted after embryos culture in vitro
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-12 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
genomic DNA in culture medium (pg) | 1 year

SECONDARY OUTCOMES:
amplification of point mutation | 1 year
  amplification of point mutation with PCR (polymerase chain reaction)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Cervesi Hospital, Cattolica
  - cervesi Hospital, Cattolica